CLINICAL TRIAL: NCT03042676
Title: Observational, Electronic Database With a Prospective Phase and Retrospective Phase for the Follow up of the ATG_FamilyStudy
Brief Title: Electronic Database for the Follow up of the ATG_FamilyStudy
Acronym: AFF
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: Universitätsklinikum Hamburg-Eppendorf (Other); Hospital Clínico Universitario de Valencia (Other); The Chaim Sheba Medical Center (Other)
Responsible Party: Principal Investigator, Francesca Bonifazi, MD, MD, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: 271/2016/O/Oss
Record Dates: First submitted 2017-01-20; First posted 2017-02-03 (Estimated); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: GVHD, Chronic; Acute Leukemia; Stem Cell Transplant Complications
Keywords: anti-T lymphocytic globulin (ATG); allogeneic stem cell transplant; prophylaxis of GVHD
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ATLG group: ATLG treatment for GVHD prophylaxis.
- no ATLG group: No ATLG treatment.

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (HSCT) is capable of definitive cure of acute leukemias. The most important post-transplant complication is graft vs host disease (GVHD) which can be substantially decreased by the addition of anti-T lymphocyte globulin (ATG-Grafalon) to the standard GVHD prophylaxis (cyclosporin and methotrexate) without any increase in relapses and infections (Kroger et al NEJM 2016, ClinicalTrials.gov number, NCT00678275). In the ATG_familystudy (prospective, randomised, multicenter study) a decrease in the incidence of chronic GVHD (from 67.8% to 32.2%) was observed after the addition of ATG (10 mg/kg for three days ,from day -3 to -1) to the standard GVHD prophylaxis in the setting of acute leukemias in any remission, receiving peripheral blood stem cells from an HLA identical sibling donor after myeloablative preparative regimen. In particular, the GVHD extensive form was reduced from 52.4% to 7.6%. The study has been closed in 2014 with a minimum follow up of 2 years from transplant. The investigators would like to evaluate the longer term follow up of this study.

DETAILED DESCRIPTION:
In the ATG_familystudy (prospective, randomised, multicenter study) a decrease in the incidence of chronic GVHD (from 67.8% to 32.2%) was observed after the addition of ATG (10 mg/kg for three days from day -3 to -1) to the standard GVHD prophylaxis in the setting of acute leukemias in any remission, receiving peripheral blood stem cells from an HLA identical sibling donor after myeloablative preparative regimen. In particular, the GVHD extensive form was reduced from 52.4% to 7.6%. The study has been closed in 2014 with a minimum follow up of 2 years from transplant.

The primary endpoint is the creation of a multicenter electronic database with data of the patients previously enrolled in the ATG_family study, NCT00678275; the data collection will last ten years. Schedule of the follow-up will have be until death and will be stopped any time if patient will retire the consent.

The database will allow to evaluate:

* Long term mortality of enrolled patients, with and without GVHD
* Long term relapse after allogeneic HSCT in acute leukemia patients
* Prognostic factors in the overall population and according to the randomization arm
* Recovery of working activity

Study design

Multicenter, observational, prospective cohorting study (electronic database) with a retrospective phase.

Prospective phase:

the electronic database will include patients enrolled in the ATG_familystudy and routinely followed up at the Hematological Institutions participating to the study.

Retrospective phase:

data collection will review all patients enrolled in the ATG familystudy (medical chart review) and already dead or lost at follow up after the end of the ATG_familystudy by medical chart review (Feb 2014).

The electronic database will include all patients enrolled in the ATG_familystudy.

Inclusion criteria:

* patients included in the ATG_familystudy (NCT00678275)
* informed consent given

Exclusion criteria: none

Treatment: no treatment is envisaged; patients are followed up according to standard clinical practice and international guidelines.

Visit and evaluation

Prospective phase: patients will be followed with visits (mainly as outpatients), laboratory and instrumental tests, phone contacts as provided for the clinic route.

Retrospective phase: medical chart review

Informed consent: patients will be asked to sign the written consent during a visit as an outpatient or inpatient, if required.

Confidentiality of collected information:

the principal investigator is the responsible of data treatment. Collected data will be analyzed by statistical methods in anonymous way in order to obtain the information representing the aim of the study. The electronic database will be accessible only by authorized persons. The principal investigator and the coworkers will have the access to data: everyone will be obliged to data confidentiality.

Electronic database

* The electronic database will include all patients enrolled in the ATG_familystudy. The data collection about hospital admittance and medical evaluations performed as outpatient will be done by medical records/charts analysis. In this way, biographical data, anamnestic data and any information about signs and symptoms at the onset of disease, diagnostic roadmap and treatment will be collected.
* For patients unreachable by phone details given by the patients or for patients already dead, data will be taken by the analysis of the medical charts or by the Office of vital statistics, after EC approval. Patients lost at follow up are patients unreachable in anyway by the details given by the patient him/herself.
* In the electronic database data on patients enrolled in the ATGfamilystudy will be included from the date of EC approval. For dead and lost at follow up patients data will be recorded retrospectively.

Statistical analysis

The investigators will use cumulative incidence analysis to assess chronic GVHD-free survival and relapse-free survival and labeled death before the event of interest as a competing risk. Death from relapse will be used as a competing risk for the cumulative incidence analysis of death without relapse. Overall survival will be assessed with the use of Kaplan- Meier analysis. Further treatment- group comparisons were performed with the use of chi-square tests for nominal data, Mann-Whitney U-tests for ordinal data, and analyses of variance for interval or ratio-scale data. Exploratory, post hoc, Cox multiple regression analysis was used for subgroup analyses and for the purpose of determining the effect on the incidence of chronic GVHD and on overall survival of recipient age, first versus second remission, acute lymphoblastic versus acute myeloid leukemia, cytogenetic risk, risk of underlying disease, difference between the sex of the donor and the sex of the recipient, cytomegalovirus positivity in the recipient, type of conditioning, CD34+ cells transplanted, grade of acute GVHD and chronic GVHD (time dependent [i.e., the corresponding event can occur at different points in time after transplantation]) in addition to treatment assignment (ATG vs. non-ATG) in the original ATG_familystudy. Confidence intervals for the differences in risk according to treatment group will be determined with the use of Wilson's method. Cumulative incidence analyses will be performed with the use of NCSS statistical software, version 9, and R statistical software, version 2.10.1 (cmprsk package). IBM SPSS Statistics software, version 22.0, will be used for all other analysis.

ELIGIBILITY:
Inclusion Criteria:

* all patients already enrolled in the ATG_family_study (NCT00678275), and published by Kroger N et al. Antilymphocyte Globulin for Prevention of Chronic Graft-versus-Host Disease. N Engl J Med 2016;374:43-53
* informed consent given

Exclusion Criteria:

* none

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The electronic database will include all patients enrolled in the ATG_familystudy (NCT00678275).
  Multicenter, observational, prospective cohorting study (electronic database) with a retrospective phase.
  Prospective phase:
  the electronic database will include patients enrolled in the ATG_familystudy and routinely followed up at the Hematological Institutions participating to the study.
  Retrospective phase:
  data collection will review all patients enrolled in the ATG familystudy (medical chart review) and already dead or lost at follow up after the end of the ATG_familystudy by medical chart review (Feb 2014)
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2018-06-08 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
cumulative incidence of cGVHD | cumulative incidence of cGVHD through study competition, an average of 24 months
  cumulative incidence according to Fine and Gray method, labeling death before the event of interest as a competing risk.

SECONDARY OUTCOMES:
Overall survival after allogeneic stem cell transplant | overall survival through study competition, an average of 24 months
  Kaplan-Meyer estimate of survival after transplant.

OTHER OUTCOMES:
Cumulative incidence of relapse after allogeneic stem cell transplant | Relapse Incidence through study competition, an average of 24 months
  cumulative incidence according to Fine and Gray method, labeling death before relapse as a competing risk.
Recovery of working activity | Recovery of working activity after transplant anytime through study competition, an average of 24 months
  descriptive measures (retired, came back to work, unemployed) during a standard follow up visit

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Bonifazi, MD, Principal Investigator — St. Orsola-Malpighi University Hospital Bologna, Italy
Locations (1):
- Hematology - Sant'Orsola-Malpighi Hospital, Bologna, Bo, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kroger N, Solano C, Wolschke C, Bandini G, Patriarca F, Pini M, Nagler A, Selleri C, Risitano A, Messina G, Bethge W, Perez de Oteiza J, Duarte R, Carella AM, Cimminiello M, Guidi S, Finke J, Mordini N, Ferra C, Sierra J, Russo D, Petrini M, Milone G, Benedetti F, Heinzelmann M, Pastore D, Jurado M, Terruzzi E, Narni F, Volp A, Ayuk F, Ruutu T, Bonifazi F. Antilymphocyte Globulin for Prevention of Chronic Graft-versus-Host Disease. N Engl J Med. 2016 Jan 7;374(1):43-53. doi: 10.1056/NEJMoa1506002. PMID 26735993
- [Result] Bonifazi F, Solano C, Wolschke C, Sessa M, Patriarca F, Zallio F, Nagler A, Selleri C, Risitano AM, Messina G, Bethge W, Herrera P, Sureda A, Carella AM, Cimminiello M, Guidi S, Finke J, Sorasio R, Ferra C, Sierra J, Russo D, Benedetti E, Milone G, Benedetti F, Heinzelmann M, Pastore D, Jurado M, Terruzzi E, Narni F, Volp A, Ayuk F, Ruutu T, Kroger N. Acute GVHD prophylaxis plus ATLG after myeloablative allogeneic haemopoietic peripheral blood stem-cell transplantation from HLA-identical siblings in patients with acute myeloid leukaemia in remission: final results of quality of life and long-term outcome analysis of a phase 3 randomised study. Lancet Haematol. 2019 Feb;6(2):e89-e99. doi: 10.1016/S2352-3026(18)30214-X. PMID 30709437